CLINICAL TRIAL: NCT00031499
Title: A Phase III Equivalence Trial of Azithromycin vs. Benzathine Penicillin for the Treatment of Early Syphilis
Brief Title: Azithromycin/Bicillin Syphilis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99-005
Record Dates: First submitted 2002-03-06; First posted 2002-03-07 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Syphilis
Keywords: Azithromycin, Syphilis, Penicillin
MeSH Terms: conditions — Syphilis | interventions — Azithromycin; Penicillin G Benzathine; Doxycycline

ARMS (2):
- Azithromycin (Experimental): Azithromycin 2.0 gram single oral dose.
  Interventions: Drug: Azithromycin
- Benzathine Penicillin (Active Comparator): Benzathine penicillin 2.4 million units administered intramuscularly. Doxycycline will be administered if the patient is allergic to Benzathine Penicillin.
  Interventions: Drug: Benzathine Penicillin; Drug: Doxycycline

INTERVENTIONS:
Drug: Azithromycin — Single 2 gram oral dose (4 tablets) at Day 1.
  Arms: Azithromycin
Drug: Benzathine Penicillin — Supplied in pre-filled syringes containing 1.2 million units of benzathine penicillin; 2.4 million units administered intramuscularly at Day 1, in one or both buttocks.
  Arms: Benzathine Penicillin
Drug: Doxycycline — Baseline visit, 28 capsules dispensed, for a dose of 100 mg twice a day (BID).
  Arms: Benzathine Penicillin

SUMMARY:
The purpose of this study is to determine if azithromycin, a drug approved for treatment of other infections, is as effective for syphilis (a sexually transmitted disease) as the standard treatment. Approximately 600 healthy adults, who are HIV-negative, ages 18 to 55 years of age, with primary, secondary or early latent syphilis, will participate in this research study. Volunteers will be enrolled in 5 U.S. cities and in Madagascar. Participants will be chosen randomly (by chance) to receive 1 of 2 study drugs: benzathine penicillin given (2 shots in the buttocks) or 4 tablets of azithromycin. Subjects who report a history of a penicillin allergy will be given either 2.0 g of oral azithromycin or 100 mg doxycycline taken orally, twice a day for 14 days. Over 2 years, 10 visits will be required. Procedures will include blood samples, physical exams, and swabs of sores.

DETAILED DESCRIPTION:
Syphilis is a disease with a worldwide distribution. It causes genital ulceration, thereby amplifying risk for HIV acquisition and transmission and it may cause congenital infection, spontaneous abortion, and stillbirth if untreated in pregnant women. About one third of all cases, if untreated, result in late sequelae which include neurosyphilis, gumma formation and cardiovascular involvement. This study will be a multi-center, randomized, open-label trial to evaluate the efficacy of azithromycin in treating primary, secondary and early latent syphilis in HIV (Human Immunodeficiency Virus) uninfected volunteers. Up through version 6.0 of this protocol volunteers were only followed for 12 months. The protocol was amended starting with version 7.0 to include follow-up visits at month 18 and 24 in order to capture possible "late failures." Each subject will be randomized into a treatment group. If the subject does not have a self-reported history of penicillin allergy, the subject will be randomized to receive either a single 2.0 gram dose of azithromycin administered orally, or 2.4 million units of benzathine penicillin G administered intramuscularly once. Eligible patients who report a history of penicillin allergy will be randomized (using a separate randomization schedule) to receive either a single dose of azithromycin or doxycycline, 100 milligrams, taken orally, twice a day for 14 days. Block randomization will be used within each clinical center with subjects allocated in equal numbers to either standard therapy or azithromycin. Participants found to be ineligible for study participation after they have been randomized and treated, will be treated again with benzathine penicillin G (or doxycycline if they are allergic to penicillin) and will continue follow-up for safety evaluation. The treatment assignments will not be blinded. No attempt will be made to recruit a sufficient sample size among penicillin allergic subjects to attain the desired power for the primary outcome. Therefore these results will be seen as preliminary to a possible future trial and as confirmatory to the primary comparison. Although the study endpoint will be determined at 6 months, all participants, will have follow-up visits for 2 full years. At the end of the 6 month evaluation period, all participants will have been classified in one of the following groups: cure; clinical response/serological nonresponse; or failure.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 to 55 years of age.
* The subject has signed written informed consent.
* The subject has untreated primary [darkfield or Treponema (T.) pallidum by a rapid, direct, fluorescent antibody darkfield (DFA-TP)] positive genital ulcers, secondary (based on classical palmar/plantar rash, condylomata lata, mucous patches, etc. or darkfield or DFA-TP positive lesions), or early latent syphilis (e.g., current reactive serologic tests for syphilis (STS), and a documented non-reactive STS or documented sexual exposure to a known early latent, primary or secondary syphilis patient in last 12 months; identification of this sexual contact must occur within 60 days of admission into the study).
* The subject has laboratory evidence of syphilis, i.e., reactive serologic test for syphilis (RPR).
* The subject is not pregnant, as documented by a negative urine or serum pregnancy test, or lactating.
* The subject is willing to have an HIV test, and, participate in HIV counseling and return to the clinic for follow-up treatment.

Exclusion Criteria:

* The subject does not have reactive serologic tests for syphilis.
* The subject has latent syphilis of unknown duration, late latent syphilis or evidence of neurosyphilis.
* The subject has a known or suspected allergy to macrolide or azalide antibiotics.
* The subject has a known or suspected sexually transmitted disease (STD), other than syphilis requiring treatment with a drug, other than azithromycin, active against T. pallidum.
* The subject has used antibiotics active against T. pallidum in the preceding 30 days. (Note: the use of antimicrobials known to NOT be effective against T. pallidum such as quinolones, sulfonamides, trimethoprim, metronidazole and spectinomycin will be allowed).
* The subject is known to be HIV positive prior to enrollment.
* The subject has suspected or known ongoing drug use that might interfere with study participation and follow-up treatment.
* The subject has a history of cardiovascular disease, known immunosuppression, or known AIDS, which might compromise response to therapy.
* The subject is judged by the investigators to be unlikely to reliably participate in the study follow-up.
* The subject has used any investigational drugs in the past 30 days.
* The subject has any other condition that may impair drug absorption (malabsorption syndrome or active peptic ulcer disease).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 593 (Actual)
Dates: Start 2000-06; Primary Completion 2007-08 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Cure of syphilis defined as a negative reactive serologic test for syphilis (RPR) titer or greater than or equal to a 4-fold (2 dilution) decrease in RPR titer at 6 months following treatment and resolution of all signs and symptoms of syphilis. | Month 6.

SECONDARY OUTCOMES:
Cure rates at 9, 12 and 24 months post treatment and the rate of relapse or reinfection defined as cure followed by recurrent clinical manifestations or a 2-dilution increase in RPR titer over previous lowest result. | Months 9, 12, and 24.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - University of Alabama Hospital - Infectious Diseases, Birmingham, Alabama
  - Indiana University, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center - Infectious Diseases, New Orleans, Louisiana
  - Johns Hopkins Hospital - Medicine - Infectious Diseases, Baltimore, Maryland
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of North Carolina School of Medicine - Center for Infectious Diseases, Chapel Hill, North Carolina
  - Durham County Health Department, Durham, North Carolina
- Madagascar (3):
  - Laboratoire National de Reference sur le VIH/SIDA (LNR), Analamanga, Antananarivo
  - Hopitaly Kely, Toamasina, Antsiranana
  - Hopitaly Mahabibo, Mahajanga Majunga, Mahajanga

REFERENCES:
- [Result] Sena AC, Wolff M, Martin DH, Behets F, Van Damme K, Leone P, Langley C, McNeil L, Hook EW. Predictors of serological cure and Serofast State after treatment in HIV-negative persons with early syphilis. Clin Infect Dis. 2011 Dec;53(11):1092-9. doi: 10.1093/cid/cir671. Epub 2011 Oct 12. PMID 21998287
- [Result] Hook EW 3rd, Behets F, Van Damme K, Ravelomanana N, Leone P, Sena AC, Martin D, Langley C, McNeil L, Wolff M. A phase III equivalence trial of azithromycin versus benzathine penicillin for treatment of early syphilis. J Infect Dis. 2010 Jun 1;201(11):1729-35. doi: 10.1086/652239. PMID 20402591